CLINICAL TRIAL: NCT06415617
Title: Effects of A Home-based Psychoeducation Programme on Subjective Well-being for Older Adults With Frailty in the Community: A Feasibility Trial
Brief Title: Home-based Psychoeducation for Older Adults With Frailty: A Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TAO An (Other)
Responsible Party: Sponsor-Investigator, TAO An, Mr, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023.585.p
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Frailty; Well-Being, Psychological
Keywords: Subjective well-being; frailty; psychoeducation
MeSH Terms: conditions — Frailty; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants will receive 60-minute weekly online group-based psychoeducation sessions for 12 weeks.
  Interventions: Other: Psychoeducation
- Control group (Active Comparator): Participants will receive 60-minute weekly online group-based physical health sessions for 12 weeks.
  Interventions: Other: Attention control

INTERVENTIONS:
Other: Psychoeducation — The content of psychoeducation is based on "Five Ways of Well-being" which covers "Be active", "Connect", "Take Notice", "Keep learning" and "Giving" . The participants will be engaged in psychoeducation through group discussion, individualised goal setting and reflective exercises.
  Arms: Experimental group
Other: Attention control — The content of the sessions mainly focuses on physical health information, such as healthy eating, physical exercise, prevention of falls, and pain management.
  Arms: Control group

SUMMARY:
This study aims to test the feasibility and acceptability of home-based psychoeducation in older adults with frailty in the community. The main questions it aims to answer are

1. Are the proposed eligibility criteria for participants and the study process in recruiting and retaining the participants appropriate?
2. Is home-based psychoeducation feasible and acceptable for older adults with frailty in the community?

Participants will receive 12 weekly online group-based sessions at their homes. The content for the experimental group and control group is different:

* Intervention group: psychoeducation
* Control group: physical health education

Participants will receive two home visits for data collection. An individual interview will be conducted with participants in the experimental group to explore their experiences.

ELIGIBILITY:
Inclusion Criteria:

(1) aged 65 years or over; (2) meeting frailty criteria by FRAIL scale (score 3 or above) ; (3) mentally competent screened by The Abbreviated Mental Test (AMT≥6) ; (4) able to speak and understand Cantonese; (5) living at home; (6) having experience using a smartphone (e.g.: sending messages, watching videos)

Exclusion Criteria:

(1) have a visual or hearing problem or a language barrier that may affect their communication or understanding; (2) being unfit for home-based exercise, as defined by having one point or above at either the 25-item Home Falls and Accidents self-reported screening tool (HOME-FAST), which is a comprehensive tool for identify home hazards for fall (3) are currently practising exercise for at least 150 minutes per week in previous four weeks; (4) are receiving active psychiatric or antidepressant treatment or joining other physical exercises or rehabilitation programmes

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Participation rate, self-reported intervention adherence, and attrition rate. | 12 weeks post-allocation
  The feasibility of the study will be measured in terms of participation rate, self-reported intervention adherence, and attrition rate.
Acceptability | 12 weeks post-allocation
  A 5-item satisfaction survey will be conducted by the end of the intervention for participants to rate the intervention in terms of appropriates of the session content, length of each session, overall intervention duration and delivery mode, from 1 (very dissatisfied) to 5 (very satisfied).

SECONDARY OUTCOMES:
Frailty level | 12 weeks post-allocation
  FRAIL scale
Physical functioning | 12 weeks post-allocation
  The Senior Fitness Test: It covers four dimensions, including muscle endurance, balance, flexibility, and tolerance measured by 30-sec arm-curl test, 30-sec chair-stand test, back-scratch test, chair sit-and-reach test, 8-foot up-and-go test, two-min step test.
Activities of daily living | 12 weeks post-allocation
  Katz Index of Independence in Activities of Daily Living
Instrumental activities of daily living | 12 weeks post-allocation
  Lawton Instrumental Activities of Daily Living Scale
Subjective well-being | 12 weeks post-allocation
  The Chinese 5-item World Health Organization Well-Being Index
Depressive symptoms | 12 weeks post-allocation
  4-item Geriatric Depression scale
Social support | 12 weeks post-allocation
  10-item Duke Social Support Index
Quality of life | 12 weeks post-allocation
  EuroQol 5-Dimension 5-Level

CONTACTS AND LOCATIONS:
Locations (1):
- The Nethersole School of Nursing, The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No